CLINICAL TRIAL: NCT06669871
Title: Effects of Weight of Dress Shirts on Arthrokinematics of Cervical Spine and Shoulders in Healthy Females Using Motion Capture Analysis: A Pilot Study
Brief Title: Effects of Weight of Dress Shirt on Arthrokinematics of Cervical Spine in Healthy Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Collaborators: Lahore University of Management Sciences (Other)
Responsible Party: Principal Investigator, Wajida Perveen, Associate Professor & Head of Physical Therapy Department, CMH Lahore Medical College and Institute of Dentistry
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 06/ERC/CMH/LMC
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Body Mass Index, Normal; Body Mass Index 18.5 or Greater
Keywords: Neck arthrokinematics;; Dress Shirt; Health females; Motion Capture Analysis

STUDY DESIGN:
Intervention Model Description: Two interventions; shirt A with customized design and another shirt B with simple design will be provided to the participants. Half of the participants will use shirt A, while remaining half will use Shirt B and their motion will be captured by hi speed cameras by trained engineers under the supervision of Co-PI. After one week of initial recording, they will be invited for second recording with the other design of the shirt.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMI-Normal (Experimental): Participants with BMI 18.50-24.50 will be included
  Interventions: Other: Shirt-A; Other: Shirt-B
- BMI greater than 25 (Experimental): Participants with BMI 25 and above will be included
  Interventions: Other: Shirt-A; Other: Shirt-B

INTERVENTIONS:
Other: Shirt-A — A dress shirt of a specific design will be provided to the participants, in which weight of the front side will be double than the back side.
Other: Shirt-B — A dress shirt of a simple design will be provided to the participants, in which weight of the front side will be equal to the back side.

SUMMARY:
Clothing is important to cover the human body, The quality of fabric is variable and a variety of designs of the dress shirts is available. Many females use biomechanically improper dress designs particularly of the shirts. This study will help us to find the effect of dress shirt design on cervical spine and shoulder joints arthrokinematics.

This non randomized pilot clinical trial with cross over assignment will be conducted on healthy female volunteers of 18-45 years of age with a BMI 18-40. Two interventions shirt with customized design will be provided to the participants. The motion will be captured by hi speed cameras by trained engineers. After one week of initial recording, participants will be invited for second recording with the other design of the shirt.

DETAILED DESCRIPTION:
Food, shelter and clothes are basic necessities of the human being. Clothing is important to cover the human body, get protected from extremes of weather, assist in one's job roles, freedom for leisure activities and for cosmetic purposes. The quality of fabric is variable and a variety of designs of the dress shirts is available. Females are about half of total population in Pakistan. Many females use biomechanically improper dress designs particularly of the shirts, which cause uneven distribution of loads to the spine and may change the angles of the individual spinal segments. This study will help us to find the effect of dress shirt design on cervical spine and shoulder joints arthrokinematics, and investigator may proceed towards designing biomechanically and ergonomically more cost effective designs in terms of mobility, energy expenditure and prevention of musculoskeletal problems. Prevention of musculoskeletal problems can have good socioeconomic impact and help in improving health outcomes in females.

This non randomized pilot clinical trial with cross over assignment will be conducted on healthy female volunteers of 18-50 years of age with a BMI 18 and above. The participants will be divided into two groups on the basis of BMI (normal and overweight). Two interventions shirt with customized design and shirt with simple design of staple Lenin fabric will be provided to the participants. Markers for motion capture will be placed on appropriate places following standard protocols. participants' motions will be captured by specific cameras by trained engineers under the supervision of Co-PI at the movement recording lab. Recording may take 5-10 minutes in one session once the participants are prepared for the procedure. After one week of initial recording, participants will be invited for second recording with the other design of the shirt. Data will be analyzed sing IBM software SPSS version 26.0. On the basis of normality of the data, parametric or non-parametric test will be selected to compute the comparative quantitative results.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years.
* BMI 18-40

Exclusion Criteria:

Females with history of cervical spine injuries. Females with history of cervical spine surgeries. Females with Congenital untreated torticollis. Females with history of shoulder complex injuries Females with recent history of tumor (spine, thorax, CA Breast, upper extremity).

Females diagnosed with osteoporosis Infection (Pulmonary and or spinal Tuberculosis). Females with Rheumatoid Arthritis. Females with Joint hyper mobility. Females unable to comply with the study protocol due to cognitive impairment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female Health volunteers
Enrollment: 16 (Actual)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
arthrokinematics of cervicle spine | With the application of intervention Shirt-A, and at 1 week with the application of intervention Shirt-B
  craniovertebral angle will be measured.

SECONDARY OUTCOMES:
recruitment of muscles on EMG | With the application of intervention Shirt-A; adopting specific static and dynamic positions , and at 1 week with the application of intervention Shirt-B, adopting specific static and dynamic positions
  Recruitment of specific muscles will be studied using surface Electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Wajida Perveen, PhD* (PT), Principal Investigator — CMH Lahore Medical College and Institute of Dentistry, Lahore Pakistan; Mian M Awais, PhD, Study Director — Lahore University of Management Sciences
Locations (1):
- School of Allied Health Sciences, CMH Lahore Medical College & Institute of Dentistry, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
only outcome specific data may be shared on reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: after completion of project and dissemination of the findings as research articles or conference papers.
Access Criteria: specific data may be shared on reasonable request to Principal Investigator.